CLINICAL TRIAL: NCT01653158
Title: A Phase 1b Dose Escalation, Open-label Study Of CP-751,871 In Combination With Docetaxel In Advanced Non-hematologic Malignancies
Brief Title: CP-751,871 In Combination With Docetaxel In Advance Non-hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021003
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Non-Hematologic Malignancies
Keywords: non-hematologic cancer; advanced solid tumors; prostrate cancer
MeSH Terms: interventions — figitumumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-751,871 combined with docetaxel (Experimental)
  Interventions: Drug: CP-751,871; Drug: Docetaxel

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 was given intravenously [IV] every 3 weeks in escalating doses ranging from 0.1 mg/kg up to 20 mg/kg.
  Standard doses of Docetaxel were given every 3 weeks with CP-751,871. Study therapy was continued until disease progression, lack of tolerability for up to 17 cycles (approximately 1 year).
Drug: Docetaxel — Docetaxel up to 75 mg/m^2 was administered intravenously [IV] on Day 1 of each 3-week dosing cycle.

SUMMARY:
This clinical trial is designed to determine the safety, tolerability, pharmacokinetics and pharmacodynamic effects of escalating doses of CP 751,871 given in combination with docetaxel in patients with non-hematologic malignancies for whom docetaxel is a reasonable treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Documented advanced-stage non-hematologic malignancy for whom docetaxel monotherapy is a reasonable treatment option
* Eastern Cooperative Oncology Group [ECOG] performance status 0-1

Exclusion Criteria:

* Significant active cardiac disease
* Chemotherapy, biological or investigational agents within 4 weeks prior to dosing
* Inadequate bone marrow, renal, cardiac or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Sutton, Surrey, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021003&StudyName=CP-751%2C871%20In%20Combination%20With%20Docetaxel%20In%20Advance%20Non-hematologic%20Malignancies

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871 0.1 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 milligram/square meter (mg/m^2) over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.1 milligram/kilogram (mg/kg) intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 0.4 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.4 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 0.8 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.8 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 1.5 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 1.5 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 3 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 3 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 6 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 6 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 10 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 10 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
- CP-751,871 20 mg/kg + Docetaxel: In the dose escalation cohort, single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously and single dose of CP-751,871 infusion 20 mg/kg intravenously were both administered on Day 1 of each cycle (1 cycle = 21 days).
  In the pharmacokinetic (PK) drug interaction expansion cohort, for Cycle 1 only, docetaxel was administered alone on Day 1 and CP-751,871 alone on Day 2; for subsequent cycles, docetaxel and CP-751,871 were both administered on Day 1.
Period: Overall Study
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Started | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 19 (Six (6) and 13 participants were enrolled in dose escalation and expansion cohorts, respectively.)
Completed | 2 | 3 | 3 | 1 | 2 | 2 | 7 | 4
Not Completed | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 15
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 9
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all enrolled participants who received single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously and single dose of CP-751,871 infusion 0.1, 0.4, 0.8, 1.5, 3, 6, 10 or 20 mg/kg intravenously at each cycle (1 cycle = 21 days).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Time Frame: Cycle 1 Day 1 through Cycle 1 Day 21
Population: Safety analysis set: all enrolled participants who started treatment, but excluding those who were enrolled in the expansion cohort.
Measure: Number; unit: mg/kg
Groups:
- CP-751,871 0.1-20 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.1, 0.4, 0.8, 1.5, 3, 6, 10 or 20 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
Arm/Group | CP-751,871 0.1-20 mg/kg + Docetaxel
Number analyzed (Participants) | 33
mg/kg | NA — Two dose limiting toxicities (DLTs) were reported (a Grade 3 fatigue, reported in a subject receiving 10 mg/kg and Grade 4 hyperglycemia reported for a subject receiving 20 mg/kg), but MTD was not reached.

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Time Frame: Cycle 1 Day 1 through Cycle 1 Day 21
Population: Safety analysis set: all enrolled participants who started treatment.
Measure: Number; unit: mg/kg
Groups:
- CP-751,871 0.1-20 mg/kg + Docetaxel: In the dose escalation cohort, single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.1, 0.4, 0.8, 1.5, 3, 6, 10 or 20 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days). In the pharmacokinetic (PK) drug interaction expansion cohort, for Cycle 1 only, docetaxel was administered alone on Day 1 and CP-751,871 alone on Day 2; for subsequent cycles, docetaxel and CP-751,871 were both administered on Day 1.
Arm/Group | CP-751,871 0.1-20 mg/kg + Docetaxel
Number analyzed (Participants) | 46
mg/kg | 20

3. Primary Outcome: Area Under the Curve From Time Zero to 25 Hours Postdose (AUC25) of Docetaxel in Cycle 1
Description: Area under the plasma concentration versus time curve (AUC) from time zero to 25 hours post dose, the nominal time of the last sample (24 hours after end of infusion)
Time Frame: 30 minutes before docetaxel infusion; 30 and 50 minutes after the start of docetaxel infusion; and 30 minutes and 1, 3, 8, and 24 hours after the end of docetaxel infusion
Population: Participants who were enrolled into the PK drug interaction expansion cohort, started treatment and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanogram*hour/millilitre (ng*hr/mL)
Groups:
- CP-751,871 20 mg/kg + Docetaxel: Cycle 1 only: single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously alone on Day 1 and single dose of CP-751,871 infusion 20 mg/kg intravenously alone on Day 2; subsequent cycles: single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 20 mg/kg intravenously on Day 1 (1 cycle = 21 days).
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
nanogram*hour/millilitre (ng*hr/mL) | 2852.11 (943.017)

4. Primary Outcome: Area Under the Curve From Time Zero to 25 Hours Postdose (AUC25) of Docetaxel in Cycle 4
Description: as for outcome 3
Time Frame: 30 minutes before CP-751,871 infusion; 1 hour after the end of CP-751,871 infusion; 30 minutes before docetaxel infusion; 30 and 50 minutes after the start of docetaxel infusion; and 30 minutes and 1, 3, 8, and 24 hours after the end of docetaxel infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
ng*hr/mL | 2526.19 (925.815)

5. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Docetaxel in Cycle 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
ng*hr/mL | 2770.71 (946.869)

6. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Docetaxel in Cycle 4
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
ng*hr/mL | 2438.34 (917.884)

7. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast(dn)) of Docetaxel in Cycle 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) divided by dose
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng•hr/mL/(mg/m^2)
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
ng•hr/mL/(mg/m^2) | 36.9428 (12.6249)

8. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast(dn)) of Docetaxel in Cycle 4
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) divided by dose
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng•hr/mL/(mg/m^2)
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
ng•hr/mL/(mg/m^2) | 35.16 (11.1288)

9. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Docetaxel in Cycle 1
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
ng/mL | 2656.92 (607.843)

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Docetaxel in Cycle 4
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
ng/mL | 2430 (497.343)

11. Primary Outcome: Dose Normalized Maximum Observed Plasma Concentration (Cmax(dn)) of Docetaxel in Cycle 1
Description: Maximum Observed Plasma Concentration (Cmax) divided by dose
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/(mg/m^2)
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
ng/mL/(mg/m^2) | 35.4256 (8.1046)

12. Primary Outcome: Dose Normalized Maximum Observed Plasma Concentration (Cmax(dn)) of Docetaxel in Cycle 4
Description: Maximum Observed Plasma Concentration (Cmax) divided by dose
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/(mg/m^2)
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
ng/mL/(mg/m^2) | 35.3 (6.0377)

13. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Docetaxel in Cycle 1
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 13
hr | 0.9179 (0.1833)

14. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Docetaxel in Cycle 4
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 5
hr | 0.8066 (0.1296)

15. Secondary Outcome: Number of Participants With the Occurrence of Human Anti-human Antibody (HAHA) Response to CP-751,871
Description: The development of HAHA is considered clinically relevant when temporally associated to the onset of adverse events or a significant decrease in the plasma concentrations of CP-751,871. The positive value is defined as ≥3.32.
Time Frame: 30 minutes predose at each cycle, End of Study (28 days after the last CP-751,871 infusion), and 150 days after the last CP-751,871 infusion
Population: All enrolled participants who started treatment and had evaluable HAHA data
Measure: Number; unit: Participants
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 3 | 3 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

16. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: Number of participants with OR based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Baseline, every 2 months (approximately 7-10 days prior to the start of the next dose) up to Cycle 17 (1 cycle = 21 days)
Population: This outcome measure was not reported because data was available in individual participant listing only and not statistically summarized for the analysis.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD])
Time Frame: as for outcome 16
Population: This outcome measure (OM) was not analyzed due to incomplete progression reporting, which could not permit accurate estimate of time to tumor progression (TTP).
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Circulating Tumor Cells (CTCs), CTCs Expressing Insulin-like Growth Factor 1 Receptor (IGF-1R), and Circulating Endothelial Cells (CECs)
Time Frame: Predose on Day 1 and on Day 8 of each cycle, and End of Study (28 days after the last CP-751,871 infusion)
Population: The data of CTCs and CTCs expressing IGF-IR were limited. Analyses of these biomarkers in the aggregate population were not feasible due to insufficient numbers. The data of CECs were not analyzed due to insufficient levels for quantification.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Systemic Clearance (CL) of CP-751,871 in Cycle 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 30 minutes prior to the Cycle 1 CP-751,871 infusion; 1 hour, and 1 (Day 2), 3 (Day 4) and 7 (Day 8) days post end of the Cycle 1 CP-751,871 infusion; and 30 minutes prior to the Cycle 2 CP-751,871 infusion (Day 22)
Population: All participants who started treatment and had evaluable PK data, excluding those who were enrolled in the PK drug interaction expansion cohort
Measure: Mean (Standard Deviation); unit: mL/day/kg
Groups:
- CP-751,871 20 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 20 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 1
mL/day/kg |  | 10.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 7.00 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 6.67 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 9.23 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. |  | 5.17 (0.99) | 3.53 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated.

20. Secondary Outcome: Systemic Clearance (CL) of CP-751,871 in Cycle 4
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 30 minutes prior to the Cycle 4 CP-751,871 infusion; 1 hour, and 1 (Day 2), 3 (Day 4) and 7 (Day 8) days post end of the Cycle 4 CP-751,871 infusion; and 30 minutes prior to the Cycle 5 CP-751,871 infusion (Day 22)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 2 | 2 | 2 | 4
mL/day/kg | 70.6 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 12.90 (0.59) | 6.84 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 3.05 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.74 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.68 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 4.01 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.70 (1.97)

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-751,871 in Cycle 1
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 6
mg/L | 1.34 (0.365) | 7.81 (0.475) | 17.9 (6.79) | 33.4 (5.97) | 57.7 (23.7) | 129 (23.6) | 205 (39.5) | 382 (156)

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-751,871 in Cycle 4
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 2 | 2 | 7 | 5
mg/L | 1.29 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 6.91 (1.75) | 17.8 (2.13) | 54.7 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 103 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 188 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 311 (65.5) | 658 (185)

23. Secondary Outcome: Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)) of CP-751,871 in Cycle 1
Description: Area under the plasma concentration versus time curve (AUC) from time zero (Day 1) to Day 22, where Day 22 is the nominal time (504 hours) of the predose sample for the next cycle.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 5
mg*hr/L | 38.4 (7.1) | 1045 (236) | 2040 (621) | 5026 (2516) | 10570 (3369) | 26215 (2520) | 38160 (7757) | 84916 (25982)

24. Secondary Outcome: Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)) of CP-751,871 in Cycle 4
Description: as for outcome 23
Time Frame: as for outcome 20
Population: This OM was not reported since the actual dosing interval (tau) was longer than 3 weeks in some patients and AUC(0-d22) may not accurately represent multiple-dose exposure for these patients. Therefore only AUCtau, which represents exposure for the actual Cycle 4 interval, was reported for Cycle 4 (OM 40).
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of CP-751,871 in Cycle 1
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 1
mg*hr/L |  | 949 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2744 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 6532 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 7799 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. |  | 47711 (9305) | 136026 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated.

26. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of CP-751,871 in Cycle 4
Description: as for outcome 25
Time Frame: as for outcome 20
Population: This OM was not reported due to registration error. AUCinf is not scientifically appropriate for repeated dosing (Cycle 4).
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CP-751,871 in Cycle 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 6
mg*hr/L | 22.3 (4.45) | 673 (127) | 1685 (879) | 4568 (2953) | 10712 (3147) | 26215 (2520) | 39724 (8380) | 78106 (37097)

28. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CP-751,871 in Cycle 4
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 2 | 2 | 7 | 5
mg*hr/L | 20.6 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 521 (37.1) | 1728 (596) | 11802 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 26329 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 55466 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 45521 (18562) | 197090 (122305)

29. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-751,871 in Cycle 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 1
hr |  | 68.5 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 97.4 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 151 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 150 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. |  | 224 (67) | 174 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated.

30. Secondary Outcome: Plasma Decay Half-Life (t1/2) of CP-751,871 in Cycle 4
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 20
Population: This OM was not reported due to insufficient data: the parameter was estimable in only 3 of 25 subjects.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CP-751,871 in Cycle 1
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 6
hr | 1.54 (0.067) | 8.76 (12.0) | 1.70 (0.146) | 9.41 (12.7) | 1.98 (0.060) | 3.21 (0.336) | 11.1 (11.5) | 8.67 (7.51)

32. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CP-751,871 in Cycle 4
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 2 | 2 | 7 | 5
hr | 1.53 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 1.65 (0.109) | 1.59 (0.119) | 2.25 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 11.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 3.23 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 9.68 (10.71) | 5.97 (0.296)

33. Secondary Outcome: Volume of Distribution at Steady State (Vss) of CP-751,871 in Cycle 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 1
mL/kg |  | 43.3 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 40.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 52.9 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 83.2 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. |  | 67.5 (15.2) | 37.5 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated.

34. Secondary Outcome: Volume of Distribution at Steady State (Vss) of CP-751,871 in Cycle 4
Description: as for outcome 33
Time Frame: as for outcome 20
Population: This OM was not reported due to insufficient data: the parameter was estimable in only 3 of 25 subjects.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of CP-751,871 in Cycle 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 19
Population: This OM was not reported due to registration error: apparent volume of distribution (Vz/F) is for oral dose. Volume of Distribution (Vz) of CP-751,871 after intravenous dosing in Cycle 1 (OM 36) was the correct outcome measure to be registered.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Volume of Distribution (Vz) of CP-751,871 in Cycle 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 1
mL/kg |  | 41.7 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 40.9 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 55.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 83.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. |  | 67.9 (15.5) | 36.8 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated.

37. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of CP-751,871 in Cycle 4
Description: as for outcome 35
Time Frame: as for outcome 20
Population: This OM was not reported due to registration error: apparent volume of distribution (Vz/F) is for oral dose. Volume of Distribution (Vz) of CP-751,871 after intravenous dosing in Cycle 4 (OM 38) was the correct outcome measure to be registered.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Volume of Distribution (Vz) of CP-751,871 in Cycle 4
Description: as for outcome 36
Time Frame: as for outcome 20
Population: This OM was not reported due to insufficient data: the parameter was estimable in only 3 of 25 subjects.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of CP-751,871 in Cycle 1
Description: Area under the plasma concentration versus time curve (AUC) from time zero to tau, the dosing interval, where tao is the actual time of the predose sample for the next cycle.
Time Frame: as for outcome 19
Population: This OM was not reported because it is the same as Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)) in Cycle 1 (OM 23), for both represented the planned 21-day dosing interval.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of CP-751,871 in Cycle 4
Description: as for outcome 39
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 2 | 2 | 2 | 4
mg*hr/L | 36.1 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 745 (34.8) | 2978 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 11802 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 26329 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 55466 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 65711 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 233578 (105208)

41. Secondary Outcome: Observed Accumulation Ratio (Rac) of CP-751,871
Description: AUCtao of Cycle 4 divided by AUC(0-d22) of Cycle 1
Time Frame: 30 minutes prior to CP-751,871 infusion; 1 hour, and 1 (Day 2), 3 (Day 4) and 7 (Day 8) days post end of CP-751,871 infusion; and 30 minutes prior to the next cycle CP-751,871 infusion (Day 22) in Cycle 1 and Cycle 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 2 | 2 | 2 | 3
Ratio | 0.852 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 0.714 (0.236) | 1.48 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 1.50 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.16 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.04 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 1.95 (NA) — Number of participants analyzed was less than 3, and thus standard deviation was not calculated. | 2.00 (0.35)

42. Other Pre Specified Outcome: Dose Normalized Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)(dn)) of CP-751,871 in Cycle 1
Description: Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)) divided by total dose
Time Frame: as for outcome 19
Population: This OM was not reported due to registration error. This parameter was not planned or analyzed for this study.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Other Pre Specified Outcome: Dose Normalized Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)(dn)) of CP-751,871 in Cycle 4
Description: Area Under the Curve From Time Zero (Day 1) to Day 22 (AUC(0-d22)) divided by total dose
Time Frame: as for outcome 20
Population: This OM was not reported due to registration error. This parameter was not planned or analyzed for this study.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Observed Concentration of CP-751,871 at Day 22 (Cday22) of Cycle 1 and 4
Description: Cday22 is the measured CP-751,871 plasma concentration in blood sample collected at Day 22.
Time Frame: Cycle 1: 30 minutes prior to the Cycle 2 CP-751,871 infusion (this is Day 22 for Cycle 1); Cycle 4: 30 minutes prior to the Cycle 5 CP-751,871 infusion (this is Day 22 for Cycle 4)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 5
mg/L
  Day 22 of Cycle 1 | 0 (0) | 0 (0) | 0.185 (0.320) | 2.11 (2.71) | 9.07 (7.17) | 30.4 (4.95) | 37.7 (15.4) | 84.5 (12.3)
  Day 22 of Cycle 4 | 0 (NA) — Number of participants analyzed was 2, which was less than 3, and thus standard deviation was not calculated. | 0 (0) | 0.144 (NA) — Number of participants analyzed was 2, which was less than 3, and thus standard deviation was not calculated. | 12.5 (NA) — Number of participants analyzed was 1, which was less than 3, and thus standard deviation was not calculated. | 32.2 (NA) — Number of participants analyzed was 2, which was less than 3, and thus standard deviation was not calculated. | 47.2 (NA) — Number of participants analyzed was 2, which was less than 3, and thus standard deviation was not calculated. | 79.3 (NA) — Number of participants analyzed was 2, which was less than 3, and thus standard deviation was not calculated. | 199 (72.9)

45. Secondary Outcome: Time of Last Quantifiable Time Point (Tlast) of CP-751,871 in Cycle 1 and Cycle 4
Description: Blood samples were collected at timepoints prespecified in the study protocol. Tlast of CP-751,871 was the last time point when blood sample collected was quantifiable for CP-751,871.
Time Frame: Cycle 1 and 4: prior to CP-751,871 infusion, at 1 hour post CP-751,871 infusion, and at 1, 3, 7 days post end of docetaxel infusion
Population: This OM was not reported due to registration error. This parameter was not planned or analyzed for this study.
Groups:
- CP-751,871 1.5 mg/kg + Docetaxel: Single dose of docetaxel infusion up to 75 mg/m^2 over 1 hour intravenously followed by single dose of CP-751,871 infusion 0.8 mg/kg intravenously on Day 1 of each cycle (1 cycle = 21 days).
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-751,871 0.1 mg/kg + Docetaxel | CP-751,871 0.4 mg/kg + Docetaxel | CP-751,871 0.8 mg/kg + Docetaxel | CP-751,871 1.5 mg/kg + Docetaxel | CP-751,871 3 mg/kg + Docetaxel | CP-751,871 6 mg/kg + Docetaxel | CP-751,871 10 mg/kg + Docetaxel | CP-751,871 20 mg/kg + Docetaxel
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 2/3 | 1/3 | 2/3 | 7/9 | 11/19
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 9/9 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 0.1 mg/kg + Docetaxel (N=3) | CP-751,871 0.4 mg/kg + Docetaxel (N=3) | CP-751,871 0.8 mg/kg + Docetaxel (N=3) | CP-751,871 1.5 mg/kg + Docetaxel (N=3) | CP-751,871 3 mg/kg + Docetaxel (N=3) | CP-751,871 6 mg/kg + Docetaxel (N=3) | CP-751,871 10 mg/kg + Docetaxel (N=9) | CP-751,871 20 mg/kg + Docetaxel (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 0.1 mg/kg + Docetaxel (N=3) | CP-751,871 0.4 mg/kg + Docetaxel (N=3) | CP-751,871 0.8 mg/kg + Docetaxel (N=3) | CP-751,871 1.5 mg/kg + Docetaxel (N=3) | CP-751,871 3 mg/kg + Docetaxel (N=3) | CP-751,871 6 mg/kg + Docetaxel (N=3) | CP-751,871 10 mg/kg + Docetaxel (N=9) | CP-751,871 20 mg/kg + Docetaxel (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 4 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 10
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 2 | 3 | 3 | 9 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 2 | 2 | 2 | 4 | 13
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 3 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 2 | 1 | 6 | 7
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Painful defaecation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 6 | 8
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 3 | 3 | 3 | 1 | 3 | 9 | 14
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 2 | 2 | 2 | 1 | 1 | 1 | 3 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Ulcer (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Blood albumin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 2
Blood glucose increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Haemoglobin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 5
White blood cell count decreased (Investigations) | 3 | 3 | 1 | 1 | 1 | 3 | 7 | 5
White blood cell count increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 2 | 2 | 5 | 7
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 3 | 3 | 2 | 2 | 1 | 5 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 2
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 4
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 4 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2 | 1 | 2 | 6 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Walking disability (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.